CLINICAL TRIAL: NCT02237014
Title: Accuracy of Peripheral Pulse Oximetry Versus Arterial Co-oximeter in Children With Cyanotic Heart Disease
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chandra Ramamoorthy, Professor, Pediatric Cardiac Anesthesia, Stanford University
Other Study IDs: SU-11062012-11219
Record Dates: First submitted 2012-11-09; First posted 2014-09-11 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Cyanotic Heart Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Peripheral pulse oximetry allows continuous non-invasive measurement of arterial oxygen saturation, but the gold standard for arterial oxygen saturation is co-oximeter which requires an arterial blood sample. The purpose of this research study is to determine the accuracy of a pulse oximeter with a standard sensor (Masimo LNCS sensor) versus with the study sensors, namely Masimo blue sensor and Nellcor Max-I sensors and compared against co-oximetry. Currently available peripheral oximeters (standard) are inaccurate at low oxygen saturation noted in children with cyanotic heart disease. Hence therapeutic interventions (including surgery and cardiac catheterizations) based solely on peripheral oximetry can be delayed and or inadequate. By doing this study the investigators will be able to establish correct limits of peripheral pulse oximeter when using the standard and the study sensors.

DETAILED DESCRIPTION:
Peripheral pulse oximetry allows continuous non-invasive measurement of arterial oxygen saturation, but the gold standard for arterial oxygen saturation is co-oximeter which requires an arterial blood sample. The purpose of this research study is to determine the accuracy of a pulse oximeter with a standard sensor (Masimo LNCS sensor) versus with the study sensors, namely Masimo blue sensor and Nellcor Max-I sensors and compared against co-oximetry. Currently available peripheral oximeters (standard) are inaccurate at low oxygen saturation noted in children with cyanotic heart disease. Hence therapeutic interventions (including surgery and cardiac catheterizations) based solely on peripheral oximetry can be delayed and or inadequate. By doing this study we will be able to establish correct limits of peripheral pulse oximeter when using the standard and the study sensors.

The investigator hopes to learn the limits of accuracy of currently available and used pulse oximeters. In children with cyanotic heart disease the "blue sensor" has been found in small studies to be more accurate compared to the "standard" pulse oximeter.

This study is important as it will provide information as to which pulse oximeter should be routinely used in children with cyanotic heart disease and to assess which SPO2 even with blue sensor is borderline and therefore the physician will know to obtain arterial blood sample for co-oximeter prior to planning important procedures based on a saturation reading.

ELIGIBILITY:
Inclusion Criteria:

1. Children from LPCH undergoing cardiac catheterization or heart surgery in SUMC or LPCH respectively
2. Peripheral arterial saturation less than or equal to 90% at time of enrollment
3. weigh between 3-20 kg
4. Less than or equal to 10 years of age

Exclusion Criteria:

1. Lack of consent
2. Greater than 10 years of age
3. Less than 3 kg or more than 20 kg in weight
4. Peripheral arterial saturation greater than 90% at time of enrollment
5. Lack of arterial access

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cyanotic heart disease undergoing cardiac catheterization or heart surgery in Stanford University Medical Center(SUMC) or Lucile Packard Children's Hospital(LPCH) respectively with peripheral arterial saturation less than 90% at time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of Peripheral Pulse Oximetry versus Arterial Co-oximeter in Children with Cyanotic Heart Disease | 2 year
  The primary outcome measure is to describe the bias and precision between the Masimo blue sensor and co-oximetry.

SECONDARY OUTCOMES:
establish correct limits of peripheral pulse oximeter when using the standard and the study sensors. | 2year
  The secondary measure was to describe the limits of the blue sensor and standard sensor accuracy as compared with the co-oximeter. If the test sensors consistently have a bias greater than 2 SD from the co-oximeter value at saturations lower than eg., 80 then the recommendation would be that the co-oximetry be used to measure patients saturatioin rather than relying on pulse oximtery alone for clinical decision making

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Ramamoorthy, MD, Principal Investigator — Department of Anesthesia, Stanford University School of Medicine
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cox P: New pulse oximetry sensors with low saturation accuracy claims-a clinical evaluation [Internet]. Anesthesiology 2007; 107:A1540
- [Background] Ross PA, Newth CJ, Khemani RG. Accuracy of pulse oximetry in children. Pediatrics. 2014 Jan;133(1):22-9. doi: 10.1542/peds.2013-1760. Epub 2013 Dec 16. PMID 24344108
- [Result] Harris BU, Char DS, Feinstein JA, Verma A, Shiboski SC, Ramamoorthy C. Accuracy of Pulse Oximeters Intended for Hypoxemic Pediatric Patients. Pediatr Crit Care Med. 2016 Apr;17(4):315-20. doi: 10.1097/PCC.0000000000000660. PMID 26914626